CLINICAL TRIAL: NCT02439762
Title: Intervening to Reduce Suicide Risk in Veterans With Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark A. Ilgen, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W81XWH 14-1-0005; Log Number 11224006 (Other Grant/Funding Number: US Army Medical Research and Materiel Command)
Record Dates: First submitted 2015-05-01; First posted 2015-05-12 (Estimated); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Suicide; Suicidal Ideation; Substance-Related Disorders
Keywords: Veterans; Cognitive Behavioral Therapy
MeSH Terms: conditions — Suicide; Suicidal Ideation; Substance-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (CBT) (Experimental): The CBT condition will cover topics such as orienting the patient to the cognitive model of suicidal thoughts, plans and behaviors and the role of substance use in increasing the likelihood of suicidal behaviors and presenting tools to help patients better manage responses to suicide-related triggers.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Supportive Psycho-education (SPC) (Active Comparator): The SPC condition is designed to match the CBT condition in terms of level of attention and the non-specific aspects of receiving support for a suicidal crisis and substance misuse. Specific content related to suicide risk will consist of general information about suicide-related resources available, while content related to substance use is based on a modified psycho-educational attention control treatment for alcoholism. The sessions will help patients to better understand the resources available during a suicidal crisis and how substance use impacts in their life. However, topics related to identifying thoughts and behaviors associated with suicidal crises and possible coping mechanisms will not be a part of the formal content of these SPC sessions.
  Interventions: Behavioral: Supportive Psycho-education (SPC)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — The therapeutic intervention group consists of 8, one-hour individual therapy sessions delivered over the course of 3-4 weeks with a trained CBT therapist. These sessions are designed to provide beneficial coping strategies that are helpful in dealing with both substance use and suicidal thoughts.
  Arms: Cognitive Behavioral Therapy (CBT)
Behavioral: Supportive Psycho-education (SPC) — This active control condition consists of 8, one-hour individual therapy sessions delivered over the course of 3-4 weeks with a trained therapist. The sessions will provide detailed information about substance use, suicide risk, and depression to those enrolled.
  Arms: Supportive Psycho-education (SPC)

SUMMARY:
The purpose of this study is to evaluate the impact of a Cognitive Behavioral Therapy (CBT) intervention compared to a Supportive Psycho-educational Control (SPC) condition in reducing the frequency and intensity of suicidal thoughts and behaviors in Veterans with Substance Use Disorders (SUDs) over a two-year follow-up period.

DETAILED DESCRIPTION:
The project is a multi-site randomized controlled trial of the CBT intervention versus the SPC condition for 300 suicidal Veterans seen in Veterans Health Administration (VHA) intensive outpatient substance treatment programs (SUD IOP). Participants will be screened for current suicidal ideation and other conditions by completing a self-report survey questionnaire. Eligible participants will complete a baseline assessment which will include a self-report survey questionnaire, a research staff administered interview, and a voluntary urine drug screen. Participants will be randomized to either a Cognitive Behavior Therapy (CBT) or Supportive Psycho-education Control (SPC) condition. Both conditions will involve receipt of 8 one-on-one sessions lasting approximately one hour over a period of approximately 3-4 weeks in addition to their standard SUD IOP treatment of care they may be receiving at the VAMC. The intervention is designed to augment their current treatment, not to take the place of current treatment. Participants will be re-assessed immediately after receiving the study interventions (at 1-month) and then again at 3-, 6- 12-, 18-, and 24-month post-intervention follow-ups by completing a series of self-report surveys, researcher administered interviews, and a voluntary urine drug screen. To ensure adequate monitoring of suicidal ideation, additional telephone follow-up assessments will occur 2-, 4-, and 5-months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Must be a United States Military Veteran
* Report current suicidal ideation
* Enrolled in outpatient substance abuse treatment within the past month
* Must live within 75 miles of treatment site at time of recruitment

Exclusion Criteria:

* Inability to give informed, voluntary, written consent
* Inability to speak and understand English
* Receipt of methadone treatment for substance use currently or within the past 6 months
* Evidence of active, severe psychotic symptoms
* Women who are currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Change in frequency and intensity of suicidal thoughts and suicide attempts | Change over study time period [Baseline, 1-, 3-, 6-, 12-, 18-, and 24-months]
  This will be measured using the Columbia Suicide Severity Rating Scale (CSS-RS) and a modified version of the Time Line Follow-Back (TLFB).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Colorado Springs, Colorado Community-Based Outpatient Clinic, Colorado Springs, Colorado
  - VA Eastern Colorado Health Care System, Denver, Colorado
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan